CLINICAL TRIAL: NCT01714609
Title: A Multi-Center, Placebo-Controlled Randomized Pilot of the Effect of Sorafenib on Portal Pressure in Patients With Cirrhosis, Portal Hypertension and Hepatocellular Carcinoma Treated With Ablative Therapy and/or Transarterial Chemoembolization
Brief Title: The Effect of Sorafenib on Portal Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002006266
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Clinically Significant Portal Hypertension
Keywords: portal hypertension; sorafenib
MeSH Terms: conditions — Hypertension, Portal | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to placebo will take two tablets of placebo by mouth twice daily.
  Interventions: Drug: Placebo
- Sorafenib (Experimental): Subjects randomized to Sorafenib will take Sorafenib 400 mg by mouth twice daily.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Placebo — Placebo Comparator: Placebo
  Arms: Placebo
Drug: Sorafenib — Sorafenib, 400 mg twice daily
  Arms: Sorafenib

SUMMARY:
Sorafenib is approved by the US FDA for the treatment of unresectable (can not operate) liver cancer and for renal cell carcinoma. Sorafenib is a drug that inhibits the growth of cancer cells and prevents the formation of new blood vessels that would otherwise help the cancer spread.

Studies in experimental animals have shown that sorafenib may also lower portal vein pressure (the pressure of the blood passing from the intestine through the liver.) This study seeks to determine if sorafenib lowers the blood pressure in liver blood vessels (portal vein pressure) in patients with cirrhosis who have high portal vein pressure. The study will also obtain information whether sorafenib is safe in this patient population.

Half of the patients will be given sorafenib and half will be given a placebo (a pill without any medicine in it.) This allows a comparison of the reactions of people who take sorafenib to those who do not.

DETAILED DESCRIPTION:
This is a pilot proof-of-concept study that investigates the effect of sorafenib on portal pressure, as determined by the hepatic venous pressure gradient (HVPG), in patients with liver cirrhosis, portal hypertension and unresectable hepatocellular carcinoma (HCC) that has successfully responded to radiofrequency ablation and/or transarterial chemoembolization, and have obtained a complete response.

The primary end-point of the study is the change in HVPG observed from baseline to three months after starting treatment with sorafenib. Secondary end-point is safety of sorafenib.

The trial is structured as a randomized double blind placebo controlled study. After a three-month period of therapy with sorafenib or placebo (double-blind phase), patients will be given open-label sorafenib for an additional 3-month period (open-label phase). A total of 44 patients will be randomized (in the initial phase) on a 1:1 ratio to sorafenib or placebo. Patients will be followed monthly and HCC follow-up will be according to standards of care. The study will be sponsored by Onyx, who will also provide the treatment medication (sorafenib and placebo)

ELIGIBILITY:
* Age 20-75 years
* Cirrhosis diagnosed by liver biopsy or by imaging studies showing a nodular liver, splenomegaly and/or collaterals
* HCC proven histologically or diagnosed following the AASLD criteria if biopsy not feasible or refused by the patient
* HCC must be unresectable and within UCSF criteria (single tumor ≤ 6.5 cm diameter, or, if multiple lesions, maximum diameter of the largest lesion ≤ 4.5 and total tumor diameter ≤ 8 cm (23))
* CPT score <9 (that is all Child A and Child B with a score of 7 or 8)
* Complete response to treatment with RFA (including that performed laparoscopically) or TACE or a combination of the above as defined by radiologic criteria (hepatoma protocol MRI or CT scan performed 4-6 weeks after the procedure).
* No more than two ablative procedures prior to enrollment
* Presence of portal hypertension, as defined by HVPG of >5 mmHg
* EGD for variceal screening performed within 6 months of entry into the study unless the patient is already on a stable dose of a non selective beta-blocker (adjusted to obtain a heart rate of 55-60 bpm) or treated with variceal band ligation.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Signed informed consent

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guadalupe Garcia-Tsao, MD, Principal Investigator — Yale University
Locations (6):
- United States (6):
  - Yale Cancer Center, New Haven, Connecticut
  - VA Medical Center West Haven, West Haven, Connecticut
  - Brigham & Womens, Boston, Massachusetts
  - New York University Langone Medical Center, New York, New York
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Sorafenib
Started | 5 | 5
Completed | 4 | 5
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sorafenib | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.98 (4.7) | 58.78 (4.25) | 57.38 (4.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Patients With Change in HVPG From Baseline
Description: Number of participants with a decrease in HPVG that was > 10% of baseline
Time Frame: Three Months
Measure: Number; unit: participants
Arm/Group | Placebo | Sorafenib
Number analyzed (Participants) | 4 | 5
participants | 1 | 1

ADVERSE EVENTS:
Description: Adverse events were collected at the organ class level, unless specified
Arm/Group | Placebo | Sorafenib
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Sorafenib (N=5)
Fever (General disorders) | 1 | 0 — Patient Hospitalized for Fever
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=5) | Sorafenib (N=5)
gastrointestinal disorders (Gastrointestinal disorders) | 5 | 5
General Disorders (General disorders) | 4 | 4
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 | 5
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3 | 2
Nervous System Disorders (Nervous system disorders) | 3 | 4
Muskoloskeletal and connective tissue (Musculoskeletal and connective tissue disorders) | 2 | 1
Psychiatric disorders (Psychiatric disorders) | 2 | 1
Respitory, thoracic and medistinal (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Vascular disorders (Vascular disorders) | 2 | 0
Alanine aminostranferase (Hepatobiliary disorders) | 1 | 0
Blood Bilirubin Increase (Hepatobiliary disorders) | 1 | 0
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 | 0
INR increased (General disorders) | 1 | 0
Infections and infestations (Infections and infestations) | 1 | 1
Platelet Count Decrease (General disorders) | 1 | 0
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 | 0
Weight Loss (Metabolism and nutrition disorders) | 1 | 1
Weight Gain (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes